CLINICAL TRIAL: NCT06712537
Title: Renal Futility Following Simultaneous Liver-Kidney Transplantation: What Identified Risk Factors to Avoid It?
Brief Title: Renal Futility Following Simultaneous Liver-Kidney Transplantation
Acronym: FUTILITY
Status: Active, not recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 24-5281
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Simultaneous Liver-kidney Transplantation
Keywords: Simultaneous liver-kidney transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Renal allograft futility: This refers to the group meeting the primary outcome, which is the need for dialysis or occurrence of death at 3 months after simultaneous liver-kidney transplantation. This group defines the absence of renal function recovery post-transplant and thus renal graft failure, termed renal futility.
- Control group

SUMMARY:
Liver transplantation in France represents a currently significant transplantation activity with a steady increase in the number of transplanted patients, with 1,294 liver transplants according to the Biomedicine Agency in 2022 compared to 806 liver transplants in 2000. 4% of these transplanted patients, or 54, underwent combined liver-kidney transplantation in 2022.

The indication for combined transplantation fits within several scenarios: patients indicated for liver transplantation with severe renal insufficiency as a comorbidity, which worsens the prognosis in the case of liver transplantation alone; patients with renal insufficiency indicated for kidney transplantation with decompensated liver disease as a comorbidity; and diseases affecting both organs in a combined and severe manner.

However, some American studies have highlighted the significant prevalence of kidney transplant failure during simultaneous liver-kidney transplantation, estimated at around 20% at 3 months post-transplant. This failure of renal function recovery after the double transplant is defined by the need for dialysis or the occurrence of death. This represents a major issue concerning the mortality and morbidity of patients who have undergone simultaneous liver-kidney transplantation.

The aim of this study is to identify the risk factors for failure of renal function recovery after combined liver-kidney transplantation, thus indicating the futility of the kidney transplant in this context of double transplantation.

The outcomes will be multiple. On one hand, we will identify the population most suitable to benefit from this intervention, which will improve recommendations on access to simultaneous liver-kidney transplantation. On the other hand, we will develop an optimized strategy for the use of available grafts, in order to better address the current organ shortage and the increasing number of patients waiting for transplants.

ELIGIBILITY:
* Inclusion Criteria * :

  * adult patient
  * having undergone simultaneous liver-kidney transplantation between January 1, 2013, and December 31, 2022
  * in France
* Exclusion Criteria * :

  * multi-organ transplant other than simultaneous liver-kidney transplantation
  * liver or kidney transplant alone
  * minor patient
  * refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects who underwent simultaneous liver-kidney transplantation between January 1, 2013, and December 31, 2022, in France
Sampling Method: Non-Probability Sample
Enrollment: 452 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Renal futility, defined as the need for dialysis (intermittent or continuous) or occurrence of death at 3 months after simultaneous liver-kidney transplantation | The outcome is collected at 3 months following the simultaneous liver-kidney transplantation.
  The primary outcome is met if the patient undergoes dialysis (continuous or intermittent) or is dead at 3 months after simultaneous liver-kidney transplantation. The outcome is not met if the patient required dialysis during the early stages of their transplant but no longer needs it and is not undergoing dialysis at 3 months. The criterion is not met if the patient dies after the 3-month period following simultaneous liver-kidney transplantation.
  This outcome is collected from electronic medical records by designated and authorized personnel. These records are stored within the hospital departments where patients are being monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Nord, HCL, Lyon, France, France